CLINICAL TRIAL: NCT03589664
Title: Computed Tomography Data Collection for Anatomical Analysis of Substernal Space in Patients With Cardiovascular Diseases
Brief Title: CT Data Collection Study
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: CT Data Collection Study
Record Dates: First submitted 2018-06-20; First posted 2018-07-18 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Cardiac Disease
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-Sternotomy Group: Subjects who have no prior sternotomy
- Sternotomy Group: Subjects who previously underwent a sternotomy procedure.

SUMMARY:
The primary objective of this study is to gather chest CT images as part of routine clinical procedure from subjects with and without prior sternotomy to characterize the substernal space. Specifically, the study will provide references for physicians to better understand substernal anatomy.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be≥18 years old
* Subject must be indicated for high quality chest CT imaging as part of routine clinical procedure
* Subject must be willing to provide Informed Consent

Exclusion Criteria:

* Subject has medical conditions that would limit study participation
* Subject is pregnant or have a pregnancy plan during the study
* Subject is enrolled in a concurrent study that may confound the results of this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll up to 100 patients who have taken or plan to take chest CT images during routine clinical procedure. The subjects will be divided into sternotomy group and non-sternotomy group based on whether the subject had undergone sternotomy.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
CT imaging data | At enrollment
  High quality CT images

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Qiu, Principal Investigator — Tongren Hospital,Shanghai Jiao Tong University School of Medicine
Locations (1):
- TongRen Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided